CLINICAL TRIAL: NCT02477670
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled, Sequential Parallel Comparison Design (SPCD) Study to Assess the Efficacy, Safety and Tolerability of AVP-786 (Deuterated [d6]-Dextromethorphan Hydrobromide [d6-DM]/Quinidine Sulfate [Q]) as an Adjunctive Treatment for Patients With Residual Schizophrenia
Brief Title: Efficacy, Safety, and Tolerability of AVP-786 for the Treatment of Residual Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Avanir Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15-AVP-786-202
Record Dates: First submitted 2015-06-18; First posted 2015-06-23 (Estimated); Results first posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-08

CONDITIONS: Schizophrenia
Keywords: Negative Symptoms; Schizophrenia; AVP-786
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo capsules administered twice a day over a 12-week period
  Interventions: Drug: Placebo
- AVP-786 (Experimental): AVP-786 dose 2 capsules administered twice a day over a 12-week period
  Interventions: Drug: AVP-786

INTERVENTIONS:
Drug: AVP-786
  Arms: AVP-786
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objectives of this 12-week study are to evaluate the efficacy, safety, and tolerability of AVP-786 as an adjunctive treatment compared with placebo in patients with residual schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet DSM-IV-TR diagnostic criteria for schizophrenia using the M.I.N.I. version 6.0.
* Patients must meet PANSS criteria
* Patients currently receiving atypical antipsychotics are eligible provided they are on a stable dose

Exclusion Criteria:

* Patients with current major depressive disorder (MDD)
* Patients with extrapyramidal syndrome secondary to their ongoing antipsychotic medication
* Patients currently using anticholinergic medications
* Recent in-patient hospitalization

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 145 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-07-21 (Actual); Study Completion 2017-07-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Cerritos, California
  - Garden Grove, California
  - National City, California
  - Oakland, California
  - San Diego, California
  - Washington D.C., District of Columbia
  - Orlando, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Chicago, Illinois
  - Boston, Massachusetts
  - Worcester, Massachusetts
  - Grand Rapids, Michigan
  - Marlton, New Jersey
  - Jamaica, New York
  - New York, New York
  - Rochester, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 145 participants randomized at the beginning of the study, 127 patients met the criteria for the Modified Intent-to-Treat (mITT) Population and were included in the Stage 1 mITT Population. A total of 108 participants were included in the Stage 2 mITT Population.
Pre-assignment Details: Participant Flow data are reported for members of the mITT Population. Stage 1: participants randomized in Stage 1 who had at least 1 post-baseline NSA-16 total score assessment in Stage 1. Stage 2: participants who were re-randomized into Stage 2 and had at least 1 NSA-16 total score assessment in Stage 2 (after Week 6).
Groups:
- Stage 1: AVP-786: Participants were randomized to receive AVP-786 once daily (QD) on Day 1 for the first 7 days. Scheduled dose escalations occurred on Day 8 and Day 14 to a target dose of AVP-786-34/4.9 milligrams twice a day (d6-DM 34 mg/Q 4.9 mg BID). Participants who completed Stage 1 were eligible to participate in Stage 2.
- Stage 1: Placebo: Participants were randomized to receive placebo capsules matched to AVP-786 orally BID. Participants who completed Stage 1 were eligible to participate in Stage 2.
- Stage 1 Placebo Non-responders; Stage 2: Placebo: Participants who were randomized to receive placebo in Stage 1 and were classified as non-responders were re-randomized to receive placebo capsules matched to AVP-786 orally BID for the entire duration of Stage 2.
- Stage 1 Placebo Non-responders; Stage 2: AVP-786: Participants who were randomized to receive placebo in Stage 1 and were classified as non-responders were re-randomized to receive AVP-786 in Stage 2 using the same dose escalation schedule used in Stage 1: AVP-786 QD on Day 1 for the first 7 days; scheduled dose escalations occurred on Day 8 and Day 14 to a target dose of AVP-786-34/4.9 BID.
- Stage 1 Placebo Responders; Stage 2: Placebo: Participants who were randomized to receive placebo in Stage 1 and were classified as responders were re-randomized to receive placebo capsules matched to AVP-786 orally BID for the entire duration of Stage 2.
- Stage 1 Placebo Responders; Stage 2: AVP-786: Participants who were randomized to receive placebo in Stage 1 and were classified as responders were re-randomized to receive AVP-786 in Stage 2 using the same dose escalation schedule used in Stage 1: AVP-786 QD on Day 1 for the first 7 days; scheduled dose escalations occurred on Day 8 and Day 14 to a target dose of AVP-786-34/4.9 BID.
- Stage 1 AVP-786; Stage 2: AVP-786: Participants who received AVP-786 in Stage 1 continued to receive AVP-786 BID in Stage 2 with no further dose escalations.
Period: Stage 1
Arm/Group | Stage 1: AVP-786 | Stage 1: Placebo | Stage 1 Placebo Non-responders; Stage 2: Placebo | Stage 1 Placebo Non-responders; Stage 2: AVP-786 | Stage 1 Placebo Responders; Stage 2: Placebo | Stage 1 Placebo Responders; Stage 2: AVP-786 | Stage 1 AVP-786; Stage 2: AVP-786
Started | 47 | 80 | 0 | 0 | 0 | 0 | 0
Completed | 43 | 67 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 13 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 7 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Non-compliance with Study Drug | 1 | 2 | 0 | 0 | 0 | 0 | 0
Period: Stage 2
Arm/Group | Stage 1: AVP-786 | Stage 1: Placebo | Stage 1 Placebo Non-responders; Stage 2: Placebo | Stage 1 Placebo Non-responders; Stage 2: AVP-786 | Stage 1 Placebo Responders; Stage 2: Placebo | Stage 1 Placebo Responders; Stage 2: AVP-786 | Stage 1 AVP-786; Stage 2: AVP-786
Started | 0 | 0 | 30 | 33 | 2 | 1 | 42
Completed | 0 | 0 | 28 | 32 | 2 | 1 | 42
Not Completed | 0 | 0 | 2 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Antipsychotic Medication Changed | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline data are reported for members of the Safety Population, comprised of all participants who received at least one dose of study medication.
Groups:
- Placebo: Participants were randomized to receive placebo capsules matched to AVP-786 orally twice a day (BID) in Stage 1.
- AVP-786: Participants were randomized to receive AVP-786 once daily (QD) on Day 1 for the first 7 days in Stage 1. Scheduled dose escalations occurred on Day 8 and Day 14 to a target dose of AVP-786-34/4.9 milligrams twice a day (d6-DM 34 mg/Q 4.9 mg BID).
- Total: Total of all reporting groups
Arm/Group | Placebo | AVP-786 | Total
Number analyzed (Participants) | 96 | 48 | 144
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.9 (10.83) | 46.5 (12.04) | 45.4 (11.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 18 | 45
  Male | 69 | 30 | 99
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 4 | 16
  Not Hispanic or Latino | 84 | 44 | 128
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 53 | 25 | 78
  White | 36 | 18 | 54
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the 16-Item Negative Symptom Assessment (NSA-16) Total Score at Week 6 and Week 12
Description: The NSA-16 is a measure of the presence, severity, and range of negative symptoms associated with schizophrenia. It has a high interrater and test-retest reliability across languages and cultures. The NSA-16 uses a 5-factor model to describe negative symptoms: (1) communication, (2) emotion/affect, (3) social involvement, (4) motivation, and (5) retardation. The possible NSA-16 total score ranges from 16 to 96, with a higher score indicating a worse condition. Change was Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Week 6 (Stage 1); Baseline (Week 6) and Week 12 (Stage 2)
Population: Modified Intent-To-Treat (mITT) Population. Stage 1: randomized participants who had at least 1 post-Baseline NSA-16 total score assessment in Stage 1. Stage 2 (Stage 1 Placebo Non-responders): re-randomized participants who had at least 1 NSA-16 total score assessment in Stage 2. Only those participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1: AVP-786 | Stage 1: Placebo | Stage 1 Placebo Non-responders; Stage 2: Placebo | Stage 1 Placebo Non-responders; Stage 2: AVP-786 | Stage 1 Placebo Responders; Stage 2: Placebo | Stage 1 Placebo Responders; Stage 2: AVP-786 | Stage 1 AVP-786; Stage 2: AVP-786
Number analyzed (Participants) | 47 | 80 | 30 | 33 | 0 | 0 | 0
score on a scale
  Stage 1 Baseline: number analyzed (Participants) | 47 | 80 | 0 | 0 | 0 | 0 | 0
  Stage 1 Baseline | 61.0 (7.53) | 60.4 (7.71) |  |  |  |  |
  Change from Baseline at Week 6: number analyzed (Participants) | 47 | 70 | 0 | 0 | 0 | 0 | 0
  Change from Baseline at Week 6 | -5.0 (5.64) | -3.4 (5.54) |  |  |  |  |
  Stage 2 Baseline: number analyzed (Participants) | 0 | 0 | 30 | 33 | 0 | 0 | 0
  Stage 2 Baseline |  |  | 57.6 (9.39) | 57.6 (9.09) |  |  |
  Change from Baseline at Week 12: number analyzed (Participants) | 0 | 0 | 29 | 32 | 0 | 0 | 0
  Change from Baseline at Week 12 |  |  | -2.4 (5.88) | -3.7 (6.41) |  |  |
Statistical Analysis 1: Comparison: Stage 1: AVP-786 vs Stage 1: Placebo vs Stage 1 Placebo Non-responders; Stage 2: Placebo vs Stage 1 Placebo Non-responders; Stage 2: AVP-786; Sequential Parallel Comparison Design (SPCD) Weighted Ordinary Least Squares (OLS) z-statistic. Treatment differences in each stage were estimated by the Mixed Model Repeated Measures (MMRM); Test type: Superiority; p = 0.073, Mixed Models Analysis; SPCD Weighted OLS z-statistic = -1.79, 95% CI 2-sided [-3.75 to 0.17]

2. Secondary Outcome: Change From Baseline in the Positive and Negative Syndrome Scale (PANSS) Total Score at Week 6 and Week 12
Description: The PANSS is a 30-item clinical scale that is extensively used as a reliable and valid measure for negative symptom trials. The PANNS consists of 6 subscales: positive subscale; negative subscale; general psychopathology subscale; prosocial factors (active social avoidance, emotional withdrawal, passive/apathetic social withdrawal, stereotyped thinking, hallucinatory behavior, suspiciousness/persecution); Marder negative factors (blunted affect, emotional withdrawal, poor rapport, passive/apathetic social withdrawal, lack of spontaneity and flow of conversation, motor retardation, active social avoidance); excitement component (excitement, hostility, tension, uncooperativeness, poor impulse control). Each item was scored from "1" (absent) to "7" (extremely severe). The PANSS total score ranges from 30 to 210, with a higher score indicating greater severity of symptoms. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Week 6 (Stage 1); Baseline (Week 6) and Week 12 (Stage 2)
Population: Stage 1 and Stage 2 mITT Populations. Only those participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1: AVP-786 | Stage 1: Placebo | Stage 1 Placebo Non-responders; Stage 2: Placebo | Stage 1 Placebo Non-responders; Stage 2: AVP-786 | Stage 1 Placebo Responders; Stage 2: Placebo | Stage 1 Placebo Responders; Stage 2: AVP-786 | Stage 1 AVP-786; Stage 2: AVP-786
Number analyzed (Participants) | 47 | 80 | 30 | 33 | 0 | 0 | 0
score on a scale
  Stage 1 Baseline: number analyzed (Participants) | 47 | 80 | 0 | 0 | 0 | 0 | 0
  Stage 1 Baseline | 67.4 (8.26) | 68.7 (7.99) |  |  |  |  |
  Change from Baseline at Week 6: number analyzed (Participants) | 47 | 70 | 0 | 0 | 0 | 0 | 0
  Change from Baseline at Week 6 | -4.7 (6.98) | -2.5 (6.50) |  |  |  |  |
  Stage 2 Baseline: number analyzed (Participants) | 0 | 0 | 30 | 33 | 0 | 0 | 0
  Stage 2 Baseline |  |  | 67.1 (9.00) | 65.6 (8.07) |  |  |
  Change from Baseline at Week 12: number analyzed (Participants) | 0 | 0 | 29 | 32 | 0 | 0 | 0
  Change from Baseline at Week 12 |  |  | -1.4 (7.64) | -4.0 (7.71) |  |  |
Statistical Analysis 1: Comparison: Stage 1: AVP-786 vs Stage 1: Placebo vs Stage 1 Placebo Non-responders; Stage 2: Placebo vs Stage 1 Placebo Non-responders; Stage 2: AVP-786; Treatment differences in each stage were estimated by the MMRM; Test type: Superiority; p = 0.025, Mixed Models Analysis; SPCD Weighted OLS z-statistic = -2.25, 95% CI 2-sided [-4.21 to -0.29]

3. Secondary Outcome: Change From Baseline in the PANSS Negative Subscale Score at Week 6 and Week 12
Description: The negative subscale includes items N1 - N7 in the PANSS. Each item was scored from "1" (absent) to "7" (extremely severe). The score ranges from 7 to 49, with higher scores indicative of greater severity of the negative symptoms. Change from Baseline was calculated as the post-Baseline score minus the Baseline score.
Time Frame: Baseline and Week 6 (Stage 1); Baseline (Week 6) and Week 12 (Stage 2)
Population: Stage 1 and Stage 2 mITT Populations. Only those participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1: AVP-786 | Stage 1: Placebo | Stage 1 Placebo Non-responders; Stage 2: Placebo | Stage 1 Placebo Non-responders; Stage 2: AVP-786 | Stage 1 Placebo Responders; Stage 2: Placebo | Stage 1 Placebo Responders; Stage 2: AVP-786 | Stage 1 AVP-786; Stage 2: AVP-786
Number analyzed (Participants) | 47 | 80 | 30 | 33 | 0 | 0 | 0
score on a scale
  Stage 1 Baseline: number analyzed (Participants) | 47 | 80 | 0 | 0 | 0 | 0 | 0
  Stage 1 Baseline | 24.6 (3.51) | 25.2 (3.64) |  |  |  |  |
  Change from Baseline at Week 6: number analyzed (Participants) | 47 | 70 | 0 | 0 | 0 | 0 | 0
  Change from Baseline at Week 6 | -2.2 (3.33) | -1.5 (3.81) |  |  |  |  |
  Stage 2 Baseline: number analyzed (Participants) | 0 | 0 | 30 | 33 | 0 | 0 | 0
  Stage 2 Baseline |  |  | 24.4 (4.55) | 23.6 (4.53) |  |  |
  Change from Baseline at Week 12: number analyzed (Participants) | 0 | 0 | 29 | 32 | 0 | 0 | 0
  Change from Baseline at Week 12 |  |  | -1.0 (2.69) | -2.3 (3.12) |  |  |
Statistical Analysis 1: Comparison: Stage 1: AVP-786 vs Stage 1: Placebo vs Stage 1 Placebo Non-responders; Stage 2: Placebo vs Stage 1 Placebo Non-responders; Stage 2: AVP-786; Treatment differences in each stage were estimated by the MMRM; Test type: Superiority; p = 0.027, Mixed Models Analysis; SPCD Weighted OLS z-statistic = -2.20, 95% CI 2-sided [-4.16 to -0.24]

4. Secondary Outcome: Change From Baseline in the PANSS Marder Negative Factor Score at Week 6 and Week 12
Description: The Marder negative factors comprise 7 items of the PANSS: N1 (blunted affect); N2 (emotional withdrawal); N3 (poor rapport); N4 (passive/apathetic social withdrawal); N6 (lack of spontaneity and flow of conversation); G7 (motor retardation), and G16 (active social avoidance). Each item is scored from "1" (absent) to "7" (extremely severe). The score ranges from 7 to 49, with higher scores indicative of greater severity of the negative symptoms of schizophrenia. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Week 6 (Stage 1); Baseline (Week 6) and Week 12 (Stage 2)
Population: Stage 1 and Stage 2 mITT Populations. Only those participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1: AVP-786 | Stage 1: Placebo | Stage 1 Placebo Non-responders; Stage 2: Placebo | Stage 1 Placebo Non-responders; Stage 2: AVP-786 | Stage 1 Placebo Responders; Stage 2: Placebo | Stage 1 Placebo Responders; Stage 2: AVP-786 | Stage 1 AVP-786; Stage 2: AVP-786
Number analyzed (Participants) | 47 | 80 | 30 | 33 | 0 | 0 | 0
score on a scale
  Stage 1 Baseline: number analyzed (Participants) | 47 | 80 | 0 | 0 | 0 | 0 | 0
  Stage 1 Baseline | 24.1 (4.24) | 24.2 (3.81) |  |  |  |  |
  Change from Baseline at Week 6: number analyzed (Participants) | 47 | 70 | 0 | 0 | 0 | 0 | 0
  Change from Baseline at Week 6 | -2.1 (3.34) | -1.6 (3.48) |  |  |  |  |
  Stage 2 Baseline: number analyzed (Participants) | 0 | 0 | 30 | 33 | 0 | 0 | 0
  Stage 2 Baseline |  |  | 23.0 (4.62) | 22.3 (5.45) |  |  |
  Change from Baseline at Week 12: number analyzed (Participants) | 0 | 0 | 29 | 32 | 0 | 0 | 0
  Change from Baseline at Week 12 |  |  | -0.8 (2.80) | -2.5 (4.27) |  |  |
Statistical Analysis 1: Comparison: Stage 1: AVP-786 vs Stage 1: Placebo vs Stage 1 Placebo Non-responders; Stage 2: Placebo vs Stage 1 Placebo Non-responders; Stage 2: AVP-786; Treatment differences in each stage were estimated by the MMRM; Test type: Superiority; p = 0.024, Mixed Models Analysis; SPCD Weighted OLS z-statistic = -2.26, 95% CI 2-sided [-4.22 to -0.3]

5. Secondary Outcome: Change From Baseline in the PANSS Prosocial Factor Subscale Score at Week 6 at Week 12
Description: The prosocial factors include items: G16 (active social avoidance); N2 (emotional withdrawal); N4 (passive/apathetic social withdrawal); N7 (stereotyped thinking); P3 (hallucinatory behavior); and P6 (suspiciousness/persecution) in the PANSS. Each item was scored from "1" (absent) to "7" (extremely severe). The score ranges from 6 to 42, with higher scores indicative of greater severity of the specific negative symptoms. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Week 6 (Stage 1); Baseline (Week 6) and Week 12 (Stage 2)
Population: Stage 1 and Stage 2 mITT Populations. Only those participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1: AVP-786 | Stage 1: Placebo | Stage 1 Placebo Non-responders; Stage 2: Placebo | Stage 1 Placebo Non-responders; Stage 2: AVP-786 | Stage 1 Placebo Responders; Stage 2: Placebo | Stage 1 Placebo Responders; Stage 2: AVP-786 | Stage 1 AVP-786; Stage 2: AVP-786
Number analyzed (Participants) | 47 | 80 | 30 | 33 | 0 | 0 | 0
score on a scale
  Stage 1 Baseline: number analyzed (Participants) | 47 | 80 | 0 | 0 | 0 | 0 | 0
  Stage 1 Baseline | 18.3 (3.24) | 18.4 (2.92) |  |  |  |  |
  Change from Baseline at Week 6: number analyzed (Participants) | 47 | 70 | 0 | 0 | 0 | 0 | 0
  Change from Baseline at Week 6 | -2.0 (2.18) | -1.1 (2.53) |  |  |  |  |
  Stage 2 Baseline: number analyzed (Participants) | 0 | 0 | 30 | 33 | 0 | 0 | 0
  Stage 2 Baseline |  |  | 17.7 (3.27) | 17.0 (3.30) |  |  |
  Change from Baseline at Week 12: number analyzed (Participants) | 0 | 0 | 29 | 32 | 0 | 0 | 0
  Change from Baseline at Week 12 |  |  | -0.7 (2.02) | -1.4 (2.35) |  |  |
Statistical Analysis 1: Comparison: Stage 1: AVP-786 vs Stage 1: Placebo vs Stage 1 Placebo Non-responders; Stage 2: Placebo vs Stage 1 Placebo Non-responders; Stage 2: AVP-786; Treatment differences in each stage were estimated by the MMRM; Test type: Superiority; p = 0.009, Mixed Models Analysis; SPCD Weighted OLS z-statistic = -2.60, 95% CI 2-sided [-4.56 to -0.64]

6. Secondary Outcome: Change From Baseline in the PANSS Positive Subscale Score at Week 6 and Week 12
Description: The positive subscale includes items P1 - P7 in the PANSS. Each item is scored from "1" (absent) to "7" (extremely severe). The score ranges from 7 to 49, with higher scores indicative of greater severity of the positive symptoms of schizophrenia. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Week 6 (Stage 1); Baseline (Week 6) and Week 12 (Stage 2)
Population: Stage 1 and Stage 2 mITT Populations. Only those participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1: AVP-786 | Stage 1: Placebo | Stage 1 Placebo Non-responders; Stage 2: Placebo | Stage 1 Placebo Non-responders; Stage 2: AVP-786 | Stage 1 Placebo Responders; Stage 2: Placebo | Stage 1 Placebo Responders; Stage 2: AVP-786 | Stage 1 AVP-786; Stage 2: AVP-786
Number analyzed (Participants) | 47 | 80 | 30 | 33 | 0 | 0 | 0
score on a scale
  Stage 1 Baseline: number analyzed (Participants) | 47 | 80 | 0 | 0 | 0 | 0 | 0
  Stage 1 Baseline | 13.6 (3.65) | 13.4 (2.81) |  |  |  |  |
  Change from Baseline at Week 6: number analyzed (Participants) | 47 | 70 | 0 | 0 | 0 | 0 | 0
  Change from Baseline at Week 6 | -0.8 (2.63) | -0.3 (2.57) |  |  |  |  |
  Stage 2 Baseline: number analyzed (Participants) | 0 | 0 | 30 | 33 | 0 | 0 | 0
  Stage 2 Baseline |  |  | 13.1 (3.64) | 13.3 (3.39) |  |  |
  Change from Baseline at Week 12: number analyzed (Participants) | 0 | 0 | 29 | 32 | 0 | 0 | 0
  Change from Baseline at Week 12 |  |  | -0.4 (1.99) | -0.3 (2.47) |  |  |
Statistical Analysis 1: Comparison: Stage 1: AVP-786 vs Stage 1: Placebo vs Stage 1 Placebo Non-responders; Stage 2: Placebo vs Stage 1 Placebo Non-responders; Stage 2: AVP-786; Treatment differences in each stage were estimated by the MMRM; Test type: Superiority; p = 0.700, Mixed Models Analysis; SPCD Weighted OLS z-statistic = -0.39, 95% CI 2-sided [-2.35 to 1.57]

7. Secondary Outcome: Change From Baseline in the PANSS General Psychopathology Subscale Score at Week 6 and Week 12
Description: The general psychopathology subscale includes items G1 - G16 in the PANSS. Each item was scored from "1" (absent) to "7" (extremely severe). The score ranges from 16 to 112, with higher scores indicative of greater severity of symptoms of schizophrenia. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Week 6 (Stage 1); Baseline (Week 6) and Week 12 (Stage 2)
Population: Stage 1 and Stage 2 mITT Populations. Only those participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1: AVP-786 | Stage 1: Placebo | Stage 1 Placebo Non-responders; Stage 2: Placebo | Stage 1 Placebo Non-responders; Stage 2: AVP-786 | Stage 1 Placebo Responders; Stage 2: Placebo | Stage 1 Placebo Responders; Stage 2: AVP-786 | Stage 1 AVP-786; Stage 2: AVP-786
Number analyzed (Participants) | 47 | 80 | 30 | 33 | 0 | 0 | 0
score on a scale
  Stage 1 Baseline: number analyzed (Participants) | 47 | 80 | 0 | 0 | 0 | 0 | 0
  Stage 1 Baseline | 29.1 (4.66) | 30.1 (5.05) |  |  |  |  |
  Change from Baseline at Week 6: number analyzed (Participants) | 47 | 70 | 0 | 0 | 0 | 0 | 0
  Change from Baseline at Week 6 | -1.7 (4.04) | -0.7 (3.21) |  |  |  |  |
  Stage 2 Baseline: number analyzed (Participants) | 0 | 0 | 30 | 33 | 0 | 0 | 0
  Stage 2 Baseline |  |  | 29.7 (5.40) | 28.7 (4.84) |  |  |
  Change from Baseline at Week 12: number analyzed (Participants) | 0 | 0 | 29 | 32 | 0 | 0 | 0
  Change from Baseline at Week 12 |  |  | 0.0 (5.14) | -1.3 (5.10) |  |  |
Statistical Analysis 1: Comparison: Stage 1: AVP-786 vs Stage 1: Placebo vs Stage 1 Placebo Non-responders; Stage 2: Placebo vs Stage 1 Placebo Non-responders; Stage 2: AVP-786; Treatment differences in each stage were estimated by the MMRM; Test type: Superiority; p = 0.054, Mixed Models Analysis; SPCD Weighted OLS z-statistic = -1.93, 95% CI 2-sided [-3.89 to 0.03]

8. Secondary Outcome: Change From Baseline in the PANSS Excitement Component Subscale Score at Week 6 and Week 12
Description: The excitement component includes items: P4 (excitement); P7 (hostility); G4 (tension); G8 (uncooperativeness); and G14 (poor impulse control). Each item is scored from "1" (absent) to "7" (extremely severe). The score ranges from 5 to 35, with higher scores indicative of greater severity of symptoms. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Week 6 (Stage 1); Baseline (Week 6) and Week 12 (Stage 2)
Population: Stage 1 and Stage 2 mITT Populations. Only those participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1: AVP-786 | Stage 1: Placebo | Stage 1 Placebo Non-responders; Stage 2: Placebo | Stage 1 Placebo Non-responders; Stage 2: AVP-786 | Stage 1 Placebo Responders; Stage 2: Placebo | Stage 1 Placebo Responders; Stage 2: AVP-786 | Stage 1 AVP-786; Stage 2: AVP-786
Number analyzed (Participants) | 47 | 80 | 30 | 33 | 0 | 0 | 0
score on a scale
  Stage 1 Baseline: number analyzed (Participants) | 47 | 80 | 0 | 0 | 0 | 0 | 0
  Stage 1 Baseline | 6.2 (1.57) | 6.3 (2.10) |  |  |  |  |
  Change from Baseline at Week 6: number analyzed (Participants) | 47 | 70 | 0 | 0 | 0 | 0 | 0
  Change from Baseline at Week 6 | -0.4 (1.64) | -0.2 (1.57) |  |  |  |  |
  Stage 2 Baseline: number analyzed (Participants) | 0 | 0 | 30 | 33 | 0 | 0 | 0
  Stage 2 Baseline |  |  | 5.8 (1.27) | 6.7 (2.59) |  |  |
  Change from Baseline at Week 12: number analyzed (Participants) | 0 | 0 | 29 | 32 | 0 | 0 | 0
  Change from Baseline at Week 12 |  |  | 0.0 (2.04) | -0.1 (1.77) |  |  |
Statistical Analysis 1: Comparison: Stage 1: AVP-786 vs Stage 1: Placebo vs Stage 1 Placebo Non-responders; Stage 2: Placebo vs Stage 1 Placebo Non-responders; Stage 2: AVP-786; Treatment differences in each stage were estimated by the MMRM; Test type: Superiority; p = 0.723, Mixed Models Analysis; SPCD Weighted OLS z-statistic = -0.35, 95% CI 2-sided [-2.31 to 1.61]

9. Secondary Outcome: Change From Baseline in the NSA-16 Communication Domain Score at Week 6 and Week 12
Description: NSA-16 Communication Factor Domain scores range from 4 to 24, with higher scores indicating greater clinical severity of symptoms. Negative values indicate improvement. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Week 6 (Stage 1); Baseline (Week 6) and Week 12 (Stage 2)
Population: Stage 1 and Stage 2 mITT Populations. Only those participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1: AVP-786 | Stage 1: Placebo | Stage 1 Placebo Non-responders; Stage 2: Placebo | Stage 1 Placebo Non-responders; Stage 2: AVP-786 | Stage 1 Placebo Responders; Stage 2: Placebo | Stage 1 Placebo Responders; Stage 2: AVP-786 | Stage 1 AVP-786; Stage 2: AVP-786
Number analyzed (Participants) | 47 | 80 | 30 | 33 | 0 | 0 | 0
score on a scale
  Stage 1 Baseline: number analyzed (Participants) | 47 | 80 | 0 | 0 | 0 | 0 | 0
  Stage 1 Baseline | 12.5 (2.54) | 12.6 (2.71) |  |  |  |  |
  Change from Baseline at Week 6: number analyzed (Participants) | 47 | 70 | 0 | 0 | 0 | 0 | 0
  Change from Baseline at Week 6 | -1.3 (2.32) | -1.0 (1.91) |  |  |  |  |
  Stage 2 Baseline: number analyzed (Participants) | 0 | 0 | 30 | 33 | 0 | 0 | 0
  Stage 2 Baseline |  |  | 12.0 (2.98) | 11.8 (3.12) |  |  |
  Change from Baseline at Week 12: number analyzed (Participants) | 0 | 0 | 29 | 32 | 0 | 0 | 0
  Change from Baseline at Week 12 |  |  | -0.4 (1.86) | -1.0 (1.56) |  |  |
Statistical Analysis 1: Comparison: Stage 1: AVP-786 vs Stage 1: Placebo vs Stage 1 Placebo Non-responders; Stage 2: Placebo vs Stage 1 Placebo Non-responders; Stage 2: AVP-786; Treatment differences in each stage were estimated by the MMRM; Test type: Superiority; p = 0.064, Mixed Models Analysis; SPCD Weighted OLS z-statistic = -1.85, 95% CI 2-sided [-3.81 to 0.11]

10. Secondary Outcome: Change From Baseline in the NSA-16 Emotion/Affect Domain Score at Week 6 and Week 12
Description: NSA-16 Emotion/Affect Domain scores range from 3 to 18, with higher scores indicating a greater clinical severity of symptoms. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Week 6 (Stage 1); Baseline (Week 6) and Week 12 (Stage 2)
Population: Stage 1 and Stage 2 mITT Populations. Only those participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1: AVP-786 | Stage 1: Placebo | Stage 1 Placebo Non-responders; Stage 2: Placebo | Stage 1 Placebo Non-responders; Stage 2: AVP-786 | Stage 1 Placebo Responders; Stage 2: Placebo | Stage 1 Placebo Responders; Stage 2: AVP-786 | Stage 1 AVP-786; Stage 2: AVP-786
Number analyzed (Participants) | 47 | 80 | 30 | 33 | 0 | 0 | 0
score on a scale
  Stage 1 Baseline: number analyzed (Participants) | 47 | 80 | 0 | 0 | 0 | 0 | 0
  Stage 1 Baseline | 12.6 (2.11) | 12.2 (1.81) |  |  |  |  |
  Change from Baseline at Week 6: number analyzed (Participants) | 47 | 70 | 0 | 0 | 0 | 0 | 0
  Change from Baseline at Week 6 | -1.0 (1.28) | -0.6 (1.54) |  |  |  |  |
  Stage 2 Baseline: number analyzed (Participants) | 0 | 0 | 30 | 33 | 0 | 0 | 0
  Stage 2 Baseline |  |  | 11.7 (1.84) | 11.7 (2.09) |  |  |
  Change from Baseline at Week 12: number analyzed (Participants) | 0 | 0 | 29 | 32 | 0 | 0 | 0
  Change from Baseline at Week 12 |  |  | -0.4 (1.50) | -0.6 (1.36) |  |  |
Statistical Analysis 1: Comparison: Stage 1: AVP-786 vs Stage 1: Placebo vs Stage 1 Placebo Non-responders; Stage 2: Placebo vs Stage 1 Placebo Non-responders; Stage 2: AVP-786; Treatment differences in each stage were estimated by the MMRM; Test type: Superiority; p = 0.100, Mixed Models Analysis; SPCD Weighted OLS z-statistic = -1.64, 95% CI 2-sided [-3.6 to 0.32]

11. Secondary Outcome: Change From Baseline in the NSA-16 Social Involvement Domain Score at Week 6 and Week 12
Description: NSA-16 Social Involvement Factor Domain scores range from 3 to 18, with higher scores indicating greater clinical severity of symptoms. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Week 6 (Stage 1); Baseline (Week 6) and Week 12 (Stage 2)
Population: Stage 1 and Stage 2 mITT Populations. Only those participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1: AVP-786 | Stage 1: Placebo | Stage 1 Placebo Non-responders; Stage 2: Placebo | Stage 1 Placebo Non-responders; Stage 2: AVP-786 | Stage 1 Placebo Responders; Stage 2: Placebo | Stage 1 Placebo Responders; Stage 2: AVP-786 | Stage 1 AVP-786; Stage 2: AVP-786
Number analyzed (Participants) | 47 | 80 | 30 | 33 | 0 | 0 | 0
score on a scale
  Stage 1 Baseline: number analyzed (Participants) | 47 | 80 | 0 | 0 | 0 | 0 | 0
  Stage 1 Baseline | 12.2 (2.02) | 12.2 (2.20) |  |  |  |  |
  Change from Baseline at Week 6: number analyzed (Participants) | 47 | 70 | 0 | 0 | 0 | 0 | 0
  Change from Baseline at Week 6 | -0.6 (1.87) | -0.3 (1.92) |  |  |  |  |
  Stage 2 Baseline: number analyzed (Participants) | 0 | 0 | 30 | 33 | 0 | 0 | 0
  Stage 2 Baseline |  |  | 12.1 (2.12) | 12.0 (2.56) |  |  |
  Change from Baseline at Week 12: number analyzed (Participants) | 0 | 0 | 29 | 32 | 0 | 0 | 0
  Change from Baseline at Week 12 |  |  | -0.8 (1.40) | -1.1 (2.51) |  |  |
Statistical Analysis 1: Comparison: Stage 1: AVP-786 vs Stage 1: Placebo vs Stage 1 Placebo Non-responders; Stage 2: Placebo vs Stage 1 Placebo Non-responders; Stage 2: AVP-786; Treatment differences in each stage were estimated by the MMRM; Test type: Superiority; p = 0.388, Mixed Models Analysis; SPCD Weighted OLS z-statistic = -0.86, 95% CI 2-sided [-2.82 to 1.1]

12. Secondary Outcome: Change From Baseline in the NSA-16 Motivation Domain Score at Week 6 and Week 12
Description: NSA-16 Motivation Factor Domain scores range from 4 to 24, with higher scores indicating greater clinical severity of symptoms. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Week 6 (Stage 1); Baseline (Week 6) and Week 12 (Stage 2)
Population: Stage 1 and Stage 2 mITT Populations. Only those participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1: AVP-786 | Stage 1: Placebo | Stage 1 Placebo Non-responders; Stage 2: Placebo | Stage 1 Placebo Non-responders; Stage 2: AVP-786 | Stage 1 Placebo Responders; Stage 2: Placebo | Stage 1 Placebo Responders; Stage 2: AVP-786 | Stage 1 AVP-786; Stage 2: AVP-786
Number analyzed (Participants) | 47 | 80 | 30 | 33 | 0 | 0 | 0
score on a scale
  Stage 1 Baseline: number analyzed (Participants) | 47 | 80 | 0 | 0 | 0 | 0 | 0
  Stage 1 Baseline | 16.5 (2.37) | 16.7 (2.33) |  |  |  |  |
  Change from Baseline at Week 6: number analyzed (Participants) | 47 | 70 | 0 | 0 | 0 | 0 | 0
  Change from Baseline at Week 6 | -1.4 (1.96) | -0.9 (1.80) |  |  |  |  |
  Stage 2 Baseline: number analyzed (Participants) | 0 | 0 | 30 | 33 | 0 | 0 | 0
  Stage 2 Baseline |  |  | 15.8 (2.61) | 15.8 (2.39) |  |  |
  Change from Baseline at Week 12: number analyzed (Participants) | 0 | 0 | 29 | 32 | 0 | 0 | 0
  Change from Baseline at Week 12 |  |  | -0.4 (2.13) | -0.4 (2.09) |  |  |
Statistical Analysis 1: Comparison: Stage 1: AVP-786 vs Stage 1: Placebo vs Stage 1 Placebo Non-responders; Stage 2: Placebo vs Stage 1 Placebo Non-responders; Stage 2: AVP-786; Treatment differences in each stage were estimated by the MMRM; Test type: Superiority; p = 0.367, Mixed Models Analysis; SPCD Weighted OLS z-statistic = -0.90, 95% CI 2-sided [-2.86 to 1.06]

13. Secondary Outcome: Change From Baseline in the NSA-16 Retardation Domain Score at Week 6 at Week 12
Description: NSA-16 Retardation Factor Domain scores range from 3 to 18, with higher scores indicating greater clinical severity of symptoms. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Week 6 (Stage 1); Baseline (Week 6) and Week 12 (Stage 2)
Population: Stage 1 and Stage 2 mITT Populations. Only those participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1: AVP-786 | Stage 1: Placebo | Stage 1 Placebo Non-responders; Stage 2: Placebo | Stage 1 Placebo Non-responders; Stage 2: AVP-786 | Stage 1 Placebo Responders; Stage 2: Placebo | Stage 1 Placebo Responders; Stage 2: AVP-786 | Stage 1 AVP-786; Stage 2: AVP-786
Number analyzed (Participants) | 47 | 80 | 30 | 33 | 0 | 0 | 0
score on a scale
  Stage 1 Baseline: number analyzed (Participants) | 47 | 80 | 0 | 0 | 0 | 0 | 0
  Stage 1 Baseline | 7.2 (1.54) | 6.7 (1.61) |  |  |  |  |
  Change from Baseline at Week 6: number analyzed (Participants) | 47 | 70 | 0 | 0 | 0 | 0 | 0
  Change from Baseline at Week 6 | -0.8 (1.46) | -0.6 (1.20) |  |  |  |  |
  Stage 2 Baseline: number analyzed (Participants) | 0 | 0 | 30 | 33 | 0 | 0 | 0
  Stage 2 Baseline |  |  | 6.0 (2.00) | 6.3 (2.05) |  |  |
  Change from Baseline at Week 12: number analyzed (Participants) | 0 | 0 | 29 | 32 | 0 | 0 | 0
  Change from Baseline at Week 12 |  |  | -0.3 (1.20) | -0.5 (1.81) |  |  |
Statistical Analysis 1: Comparison: Stage 1: AVP-786 vs Stage 1: Placebo vs Stage 1 Placebo Non-responders; Stage 2: Placebo vs Stage 1 Placebo Non-responders; Stage 2: AVP-786; Treatment differences in each stage were estimated by the MMRM; Test type: Superiority; p = 0.447, Mixed Models Analysis; SPCD Weighted OLS z-statistic = -0.76, 95% CI 2-sided [-2.72 to 1.2]

14. Secondary Outcome: Change From Baseline in the NSA-16 Global Negative Symptoms Score at Week 6 and Week 12
Description: The global negative symptoms rating in the NSA-16 is a single score based on the overall impression of severity of negative symptoms on a 1 to 7 scale, where higher scores indicate greater severity. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Week 6 (Stage 1); Baseline (Week 6) and Week 12 (Stage 2)
Population: Stage 1 and Stage 2 mITT Populations. Only those participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1: AVP-786 | Stage 1: Placebo | Stage 1 Placebo Non-responders; Stage 2: Placebo | Stage 1 Placebo Non-responders; Stage 2: AVP-786 | Stage 1 Placebo Responders; Stage 2: Placebo | Stage 1 Placebo Responders; Stage 2: AVP-786 | Stage 1 AVP-786; Stage 2: AVP-786
Number analyzed (Participants) | 47 | 80 | 30 | 33 | 0 | 0 | 0
score on a scale
  Stage 1 Baseline: number analyzed (Participants) | 47 | 80 | 0 | 0 | 0 | 0 | 0
  Stage 1 Baseline | 4.6 (0.64) | 4.6 (0.61) |  |  |  |  |
  Change from Baseline at Week 6: number analyzed (Participants) | 47 | 70 | 0 | 0 | 0 | 0 | 0
  Change from Baseline at Week 6 | -0.4 (0.68) | -0.2 (0.64) |  |  |  |  |
  Stage 2 Baseline: number analyzed (Participants) | 0 | 0 | 30 | 33 | 0 | 0 | 0
  Stage 2 Baseline |  |  | 4.3 (0.71) | 4.4 (0.75) |  |  |
  Change from Baseline at Week 12: number analyzed (Participants) | 0 | 0 | 29 | 32 | 0 | 0 | 0
  Change from Baseline at Week 12 |  |  | -0.1 (0.51) | -0.5 (0.75) |  |  |
Statistical Analysis 1: Comparison: Stage 1: AVP-786 vs Stage 1: Placebo vs Stage 1 Placebo Non-responders; Stage 2: Placebo vs Stage 1 Placebo Non-responders; Stage 2: AVP-786; Treatment differences in each stage were estimated by the MMRM; Test type: Superiority; p = 0.026, Mixed Models Analysis; SPCD Weighted OLS z-statistic = -2.23, 95% CI 2-sided [-4.19 to -0.27]

15. Secondary Outcome: Change From Baseline in the NSA-16 Global Level of Functioning Score at Week 6 and Week 12
Description: The global level of functioning is a single score on a scale of 1 to 7 that provides the overall assessment of the participant's level of functioning, with higher scores indicative of severe impairment in functioning. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Week 6 (Stage 1); Baseline (Week 6) and Week 12 (Stage 2)
Population: Stage 1 and Stage 2 mITT Populations. Only those participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1: AVP-786 | Stage 1: Placebo | Stage 1 Placebo Non-responders; Stage 2: Placebo | Stage 1 Placebo Non-responders; Stage 2: AVP-786 | Stage 1 Placebo Responders; Stage 2: Placebo | Stage 1 Placebo Responders; Stage 2: AVP-786 | Stage 1 AVP-786; Stage 2: AVP-786
Number analyzed (Participants) | 46 | 80 | 29 | 33 | 0 | 0 | 0
score on a scale
  Stage 1 Baseline: number analyzed (Participants) | 46 | 80 | 0 | 0 | 0 | 0 | 0
  Stage 1 Baseline | 4.7 (0.73) | 4.6 (0.63) |  |  |  |  |
  Change from Baseline at Week 6: number analyzed (Participants) | 46 | 80 | 0 | 0 | 0 | 0 | 0
  Change from Baseline at Week 6 | -0.4 (0.61) | -0.2 (0.55) |  |  |  |  |
  Stage 2 Baseline: number analyzed (Participants) | 0 | 0 | 29 | 33 | 0 | 0 | 0
  Stage 2 Baseline |  |  | 4.5 (0.74) | 4.4 (0.70) |  |  |
  Change from Baseline at Week 12: number analyzed (Participants) | 0 | 0 | 28 | 32 | 0 | 0 | 0
  Change from Baseline at Week 12 |  |  | -0.3 (0.52) | -0.3 (0.64) |  |  |
Statistical Analysis 1: Comparison: Stage 1: AVP-786 vs Stage 1: Placebo vs Stage 1 Placebo Non-responders; Stage 2: Placebo vs Stage 1 Placebo Non-responders; Stage 2: AVP-786; Treatment differences in each stage were estimated by the MMRM; Test type: Superiority; p = 0.106, Mixed Models Analysis; SPCD Weighted OLS z-statistic = -1.62, 95% CI 2-sided [-3.58 to 0.34]

16. Secondary Outcome: Change From Baseline in the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB) Composite Score at Week 6 and Week 12
Description: The MCCB is the standard tool for assessing cognitive change in trials of cognitive-enhancing agents in schizophrenia and is used to provide a relatively brief evaluation of key cognitive domains relevant to schizophrenia and related disorders. It is made up of 10 tests that measure 7 cognitive domains: Speed of Processing; Attention/Vigilance; Working Memory; Verbal Learning; Visual Learning; Reasoning and Problem Solving; and Social Cognition. The MCCB was to be conducted at approximately the same time of day (+/- 2 hours) and preferably in the morning. The MCCB composite score ranges from 0 to 70, with higher scores indicative of less severe cognition symptoms. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Week 6 (Stage 1); Baseline (Week 6) and Week 12 (Stage 2)
Population: Stage 1 and Stage 2 mITT Populations. Only those participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1: AVP-786 | Stage 1: Placebo | Stage 1 Placebo Non-responders; Stage 2: Placebo | Stage 1 Placebo Non-responders; Stage 2: AVP-786 | Stage 1 Placebo Responders; Stage 2: Placebo | Stage 1 Placebo Responders; Stage 2: AVP-786 | Stage 1 AVP-786; Stage 2: AVP-786
Number analyzed (Participants) | 47 | 80 | 30 | 33 | 0 | 0 | 0
score on a scale
  Stage 1 Baseline: number analyzed (Participants) | 47 | 80 | 0 | 0 | 0 | 0 | 0
  Stage 1 Baseline | 32.5 (11.37) | 28.8 (13.09) |  |  |  |  |
  Change from Baseline at Week 6: number analyzed (Participants) | 46 | 75 | 0 | 0 | 0 | 0 | 0
  Change from Baseline at Week 6 | 1.2 (5.11) | 1.6 (4.55) |  |  |  |  |
  Stage 2 Baseline: number analyzed (Participants) | 0 | 0 | 30 | 33 | 0 | 0 | 0
  Stage 2 Baseline |  |  | 31.7 (14.99) | 28.9 (10.69) |  |  |
  Change from Baseline at Week 12: number analyzed (Participants) | 0 | 0 | 27 | 30 | 0 | 0 | 0
  Change from Baseline at Week 12 |  |  | -1.6 (4.06) | 1.6 (3.71) |  |  |
Statistical Analysis 1: Comparison: Stage 1: AVP-786 vs Stage 1: Placebo vs Stage 1 Placebo Non-responders; Stage 2: Placebo vs Stage 1 Placebo Non-responders; Stage 2: AVP-786; Treatment differences in each stage were estimated by the MMRM; Test type: Superiority; p = 0.074, Mixed Models Analysis; SPCD Weighted OLS z-statistic = 1.78, 95% CI 2-sided [-0.18 to 3.74]

17. Secondary Outcome: Mean Actual Clinical Global Impression of Severity (CGI-S) of Illness Score at Week 6 and Week 12
Description: The CGI is an assessment of a participant's global functioning prior to and after initiating study medication and provides an overall clinician-determined summary measure that takes into account knowledge of the participant's history, psychosocial circumstances, symptoms, behavior, and the impact of the symptoms on the participant's ability to function. It is based on a 7-point scale that requires the clinician to rate the severity of the participant's illness at the time of assessment, relative to the clinician's past experience with participants who have the same diagnosis. Considering the total clinical experience, a participant is assessed on severity of mental illness at the time of rating: 1 (normal, not at all ill); 2 (borderline mentally ill); 3 (mildly ill); 4 (moderately ill); 5 (markedly ill); 6 (severely ill); or 7 (among the most extremely ill participants). Scores range from 1 to 7, with higher scores indicative of greater severity of illness.
Time Frame: Week 6 (Stage 1); Week 12 (Stage 2)
Population: Stage 1 and Stage 2 mITT Populations. Only those participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1: AVP-786 | Stage 1: Placebo | Stage 1 Placebo Non-responders; Stage 2: Placebo | Stage 1 Placebo Non-responders; Stage 2: AVP-786 | Stage 1 Placebo Responders; Stage 2: Placebo | Stage 1 Placebo Responders; Stage 2: AVP-786 | Stage 1 AVP-786; Stage 2: AVP-786
Number analyzed (Participants) | 46 | 78 | 30 | 31 | 0 | 0 | 0
score on a scale
  Week 6: number analyzed (Participants) | 46 | 78 | 0 | 0 | 0 | 0 | 0
  Week 6 | 3.6 (0.80) | 3.8 (0.77) |  |  |  |  |
  Week 12: number analyzed (Participants) | 0 | 0 | 30 | 31 | 0 | 0 | 0
  Week 12 |  |  | 3.7 (0.75) | 3.5 (0.93) |  |  |
Statistical Analysis 1: Comparison: Stage 1: AVP-786 vs Stage 1: Placebo vs Stage 1 Placebo Non-responders; Stage 2: Placebo vs Stage 1 Placebo Non-responders; Stage 2: AVP-786; Treatment differences in each stage were estimated by the MMRM; Test type: Superiority; p = 0.427, Mixed Models Analysis; SPCD Weighted OLS z-statistic = -0.79, 95% CI 2-sided [-2.75 to 1.17]

18. Secondary Outcome: Mean Actual Clinical Global Impression of Change (CGI-C) Score at Week 6 and Week 12
Description: The CGI is an assessment of the participant's global functioning prior to and after initiating a study medication and provides an overall clinician-determined summary measure that takes into account all available information, including knowledge of the participant's history, psychosocial circumstances, symptoms, behavior, and the impact of the symptoms on the participant's ability to function. It is based on a 7-point scale that requires the clinician to rate the change of the participant's condition at the time of assessment, relative to the clinician's past experience with the participant's condition at admission. Considering the total clinical experienced, a participant is assessed for change of mental illness as: 1 (very much improved); 2 (much improved); 3 (minimally improved); 4 (no change); 5 (minimally worse); 6 (much worse); or 7 (very much worse). Scores range from 1 to 7, with higher scores indicative of greater severity of illness.
Time Frame: Baseline, Week 6 (Stage 1), Week 12 (Stage 2)
Population: Stage 1 and Stage 2 mITT Populations. Only those participants with available data were analyzed. Week 6 scores are relative to Stage 1 Baseline. Week 12 scores are relative to Week 6.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1: AVP-786 | Stage 1: Placebo | Stage 1 Placebo Non-responders; Stage 2: Placebo | Stage 1 Placebo Non-responders; Stage 2: AVP-786 | Stage 1 Placebo Responders; Stage 2: Placebo | Stage 1 Placebo Responders; Stage 2: AVP-786 | Stage 1 AVP-786; Stage 2: AVP-786
Number analyzed (Participants) | 47 | 78 | 30 | 32 | 0 | 0 | 0
score on a scale
  Week 6: number analyzed (Participants) | 47 | 78 | 0 | 0 | 0 | 0 | 0
  Week 6 | 3.4 (0.80) | 3.6 (0.69) |  |  |  |  |
  Week 12: number analyzed (Participants) | 0 | 0 | 30 | 32 | 0 | 0 | 0
  Week 12 |  |  | 3.8 (0.90) | 3.5 (0.80) |  |  |
Statistical Analysis 1: Comparison: Stage 1: AVP-786 vs Stage 1: Placebo vs Stage 1 Placebo Non-responders; Stage 2: Placebo vs Stage 1 Placebo Non-responders; Stage 2: AVP-786; Treatment differences in each stage were estimated by the MMRM; Test type: Superiority; p = 0.0566, McNemar; SPCD Weighted OLS z-statistic = -1.91, 95% CI 2-sided [-3.87 to 0.05]

19. Secondary Outcome: Mean Actual Patient Global Impression of Change (PGI-C) Score at Week 6 at Week 12
Description: The PGI-C is a 7-point, participant-rated scale used to assess treatment response as: 0=Not assessed; 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally 6=worse; or 7=very much worse. Week 6 and Week 12 scores are relative to Stage 1 Baseline.
Time Frame: Baseline, Week 6 (Stage 1), Week 12 (Stage 2)
Population: Stage 1 and Stage 2 mITT Populations. Only those participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1: AVP-786 | Stage 1: Placebo | Stage 1 Placebo Non-responders; Stage 2: Placebo | Stage 1 Placebo Non-responders; Stage 2: AVP-786 | Stage 1 Placebo Responders; Stage 2: Placebo | Stage 1 Placebo Responders; Stage 2: AVP-786 | Stage 1 AVP-786; Stage 2: AVP-786
Number analyzed (Participants) | 47 | 75 | 30 | 32 | 0 | 0 | 0
score on a scale
  Week 6: number analyzed (Participants) | 47 | 75 | 0 | 0 | 0 | 0 | 0
  Week 6 | 3.1 (0.94) | 3.2 (1.01) |  |  |  |  |
  Week 12: number analyzed (Participants) | 0 | 0 | 30 | 32 | 0 | 0 | 0
  Week 12 |  |  | 3.3 (0.78) | 2.9 (1.11) |  |  |
Statistical Analysis 1: Comparison: Stage 1: AVP-786 vs Stage 1: Placebo vs Stage 1 Placebo Non-responders; Stage 2: Placebo vs Stage 1 Placebo Non-responders; Stage 2: AVP-786; Test type: Superiority; p = 0.1700, ANCOVA; SPCD Weighted OLS z-statistic = -1.37, 95% CI 2-sided [-3.33 to 0.59]

20. Secondary Outcome: Change From Baseline in the Calgary Depression Scale for Schizophrenia (CDSS) Total Score at Week 6 and Week 12
Description: The CDSS is a 9-item scale derived from the Hamilton Depression Scale (Ham-D) that is designed to assess depression specifically in participants with schizophrenia. Unlike the Ham-D, the CDSS does not contain depressive symptoms that overlap with negative symptoms of schizophrenia, such as anhedonia and social withdrawal. Each item on the scale is scored as: 0 (absent); 1 (mild); 2 (moderate); or 3 (severe). The CDSS is obtained by adding each of the item scores. A score above 6 has an 82% specificity and 85% sensitivity for predicting the presence of a major depressive episode. The CDSS score ranges from 0 to 27, with higher scores indicative of severe symptoms of depression. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Week 6 (Stage 1); Baseline (Week 6) and Week 12 (Stage 2)
Population: Stage 1 and Stage 2 mITT Populations. Only those participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1: AVP-786 | Stage 1: Placebo | Stage 1 Placebo Non-responders; Stage 2: Placebo | Stage 1 Placebo Non-responders; Stage 2: AVP-786 | Stage 1 Placebo Responders; Stage 2: Placebo | Stage 1 Placebo Responders; Stage 2: AVP-786 | Stage 1 AVP-786; Stage 2: AVP-786
Number analyzed (Participants) | 47 | 80 | 30 | 33 | 0 | 0 | 0
score on a scale
  Stage 1 Baseline: number analyzed (Participants) | 47 | 80 | 0 | 0 | 0 | 0 | 0
  Stage 1 Baseline | 1.1 (1.34) | 0.9 (1.31) |  |  |  |  |
  Chane from Baseline at Week 6: number analyzed (Participants) | 47 | 70 | 0 | 0 | 0 | 0 | 0
  Chane from Baseline at Week 6 | -0.2 (1.34) | -0.1 (1.02) |  |  |  |  |
  Stage 2 Baseline: number analyzed (Participants) | 0 | 0 | 30 | 33 | 0 | 0 | 0
  Stage 2 Baseline |  |  | 1.0 (1.56) | 0.8 (1.54) |  |  |
  Change from Baseline at Week 12: number analyzed (Participants) | 0 | 0 | 29 | 32 | 0 | 0 | 0
  Change from Baseline at Week 12 |  |  | -0.4 (1.24) | -0.0 (1.66) |  |  |
Statistical Analysis 1: Comparison: Stage 1: AVP-786 vs Stage 1: Placebo vs Stage 1 Placebo Non-responders; Stage 2: Placebo vs Stage 1 Placebo Non-responders; Stage 2: AVP-786; Treatment differences in each stage were estimated by the MMRM; Test type: Superiority; p = 0.595, Mixed Models Analysis; SPCD Weighted OLS z-statistic = 0.53, 95% CI 2-sided [-1.43 to 2.49]

21. Secondary Outcome: Change From Baseline in the Effort Expenditure for Reward Task (EEfRT) Score for Baseline Press Rate at Week 6 and Week 12
Description: The EEfRT is a multi-trial computerized task in which participants are given the opportunity on each trial to choose between 2 tasks that differ in difficulty level and are associated with varying levels of monetary reward. The test measures drug effects on the willingness to expend effort in relation to the amount of reward or probability of reward. The ratio of hard task choices with moderate probability reward is used as an outcome measure for negative symptoms. EEfRT scores are analyzed for 8 variables. Variable 1 is the Baseline press rate and is defined as the value coded as average presses/second. Scores range from 0 to 9, with higher scores indicative of faster button pressing ability. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Week 6 (Stage 1); Baseline (Week 6) and Week 12 (Stage 2)
Population: Stage 1 and Stage 2 mITT Populations. Only those participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1: AVP-786 | Stage 1: Placebo | Stage 1 Placebo Non-responders; Stage 2: Placebo | Stage 1 Placebo Non-responders; Stage 2: AVP-786 | Stage 1 Placebo Responders; Stage 2: Placebo | Stage 1 Placebo Responders; Stage 2: AVP-786 | Stage 1 AVP-786; Stage 2: AVP-786
Number analyzed (Participants) | 42 | 66 | 18 | 25 | 0 | 0 | 0
score on a scale
  Stage 1 Baseline: number analyzed (Participants) | 42 | 66 | 0 | 0 | 0 | 0 | 0
  Stage 1 Baseline | 3.39 (1.137) | 3.39 (1.112) |  |  |  |  |
  Change from Baseline at Week 6: number analyzed (Participants) | 38 | 49 | 0 | 0 | 0 | 0 | 0
  Change from Baseline at Week 6 | 0.461 (0.844) | 0.195 (1.181) |  |  |  |  |
  Stage 2 Baseline: number analyzed (Participants) | 0 | 0 | 18 | 25 | 0 | 0 | 0
  Stage 2 Baseline |  |  | 3.38 (1.284) | 3.67 (0.904) |  |  |
  Change from Baseline at Week 12: number analyzed (Participants) | 0 | 0 | 18 | 25 | 0 | 0 | 0
  Change from Baseline at Week 12 |  |  | -0.109 (0.909) | 0.354 (1.076) |  |  |
Statistical Analysis 1: Comparison: Stage 1: AVP-786 vs Stage 1: Placebo vs Stage 1 Placebo Non-responders; Stage 2: Placebo vs Stage 1 Placebo Non-responders; Stage 2: AVP-786; Test type: Superiority; p = 0.022, ANCOVA; SPCD Weighted OLS z-statistic = 2.284, 95% CI 2-sided [0.324 to 4.244]

22. Secondary Outcome: Change From Baseline in the EEfRT Score for Choice Reaction Time (RT) 1st 50 at Week 6 and Week 12
Description: The EEfRT is a multi-trial computerized test that reliably measures drug effects on the willingness to expend effort in relation to the amount of reward or probability of reward. For each trial, participants are asked to choose between 2 tasks that differ in difficulty level and are associated with varying levels of monetary reward. EEfRT scores are analyzed for 8 variables. Variable 2 is the choice RT and is defined as the average RT measured in milliseconds for making a choice during the first 50 trials. Scores range from 0 to 10,000. The target range is greater than 500. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Week 6 (Stage 1); Baseline (Week 6) and Week 12 (Stage 2)
Population: Stage 1 and Stage 2 mITT Populations. Only those participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1: AVP-786 | Stage 1: Placebo | Stage 1 Placebo Non-responders; Stage 2: Placebo | Stage 1 Placebo Non-responders; Stage 2: AVP-786 | Stage 1 Placebo Responders; Stage 2: Placebo | Stage 1 Placebo Responders; Stage 2: AVP-786 | Stage 1 AVP-786; Stage 2: AVP-786
Number analyzed (Participants) | 42 | 65 | 18 | 25 | 0 | 0 | 0
score on a scale
  Stage 1 Baseline: number analyzed (Participants) | 42 | 65 | 0 | 0 | 0 | 0 | 0
  Stage 1 Baseline | 1339.5 (838.40) | 1659.4 (1063.02) |  |  |  |  |
  Change from Baseline at Week 6: number analyzed (Participants) | 39 | 50 | 0 | 0 | 0 | 0 | 0
  Change from Baseline at Week 6 | -255.1 (551.65) | -346.6 (1108.63) |  |  |  |  |
  Stage 2 Baseline: number analyzed (Participants) | 0 | 0 | 18 | 25 | 0 | 0 | 0
  Stage 2 Baseline |  |  | 1309.4 (595.02) | 1283.5 (875.79) |  |  |
  Change from Baseline at Week 12: number analyzed (Participants) | 0 | 0 | 18 | 25 | 0 | 0 | 0
  Change from Baseline at Week 12 |  |  | -288.8 (527.42) | -110.2 (812.66) |  |  |
Statistical Analysis 1: Comparison: Stage 1: AVP-786 vs Stage 1: Placebo vs Stage 1 Placebo Non-responders; Stage 2: Placebo vs Stage 1 Placebo Non-responders; Stage 2: AVP-786; Test type: Superiority; p = 0.862, ANCOVA; SPCD Weighted OLS z-statistic = -0.17, 95% CI 2-sided [-2.13 to 1.79]

23. Secondary Outcome: Change From Baseline in the EEfRT Score for Completed Tasks at Week 6 and Week 12
Description: The EEfRT is a multi-trial computerized test that reliably measures drug effects on the willingness to expend effort in relation to the amount of reward or probability of reward. For each trial, participants are asked to choose between 2 tasks that differ in difficulty level and are associated with varying levels of monetary reward. EEfRT scores are analyzed for 8 variables. Variable 3 is the proportion of completed task (easy or hard) during the first 50 trials. Scores range from 0 to 1, with higher scores indicative of better task compliance. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Week 6 (Stage 1); Baseline (Week 6) and Week 12 (Stage 2)
Population: Stage 1 and Stage 2 mITT Populations. Only those participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1: AVP-786 | Stage 1: Placebo | Stage 1 Placebo Non-responders; Stage 2: Placebo | Stage 1 Placebo Non-responders; Stage 2: AVP-786 | Stage 1 Placebo Responders; Stage 2: Placebo | Stage 1 Placebo Responders; Stage 2: AVP-786 | Stage 1 AVP-786; Stage 2: AVP-786
Number analyzed (Participants) | 42 | 66 | 18 | 25 | 0 | 0 | 0
score on a scale
  Stage 1 Baseline: number analyzed (Participants) | 42 | 66 | 0 | 0 | 0 | 0 | 0
  Stage 1 Baseline | 0.790 (0.285) | 0.749 (0.294) |  |  |  |  |
  Change from Baseline at Week 6: number analyzed (Participants) | 39 | 50 | 0 | 0 | 0 | 0 | 0
  Change from Baseline at Week 6 | -0.032 (0.196) | 0.001 (0.209) |  |  |  |  |
  Stage 2 Baseline: number analyzed (Participants) | 0 | 0 | 18 | 25 | 0 | 0 | 0
  Stage 2 Baseline |  |  | 0.703 (0.329) | 0.779 (0.254) |  |  |
  Change from Baseline at Week 12: number analyzed (Participants) | 0 | 0 | 18 | 25 | 0 | 0 | 0
  Change from Baseline at Week 12 |  |  | 0.049 (0.223) | -0.022 (0.173) |  |  |
Statistical Analysis 1: Comparison: Stage 1: AVP-786 vs Stage 1: Placebo vs Stage 1 Placebo Non-responders; Stage 2: Placebo vs Stage 1 Placebo Non-responders; Stage 2: AVP-786; Test type: Superiority; p = 0.251, ANCOVA; SPCD Weighted OLS z-statistic = -1.149, 95% CI 2-sided [-3.109 to 0.811]

24. Secondary Outcome: Change From Baseline in the EEfRT Score for 12% Probability-Proportion High Effort Opts at Week 6 and Week 12
Description: The EEfRT is a multi-trial computerized test that reliably measures drug effects on the willingness to expend effort in relation to the amount of reward or probability of reward. For each trial, participants are asked to choose between 2 tasks that differ in difficulty level and are associated with varying levels of monetary reward. EEfRT scores are analyzed for 8 variables. Variable 4 is the proportion of hard task choices made for the low (12%) probability condition during the first 50 trials of the task. Scores range from 0 to 1, with higher scores indicative of greater effort expenditure. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Week 6 (Stage 1); Baseline (Week 6) and Week 12 (Stage 2)
Population: Stage 1 and Stage 2 mITT Populations. Only those participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1: AVP-786 | Stage 1: Placebo | Stage 1 Placebo Non-responders; Stage 2: Placebo | Stage 1 Placebo Non-responders; Stage 2: AVP-786 | Stage 1 Placebo Responders; Stage 2: Placebo | Stage 1 Placebo Responders; Stage 2: AVP-786 | Stage 1 AVP-786; Stage 2: AVP-786
Number analyzed (Participants) | 42 | 65 | 17 | 25 | 0 | 0 | 0
score on a scale
  Stage 1 Baseline: number analyzed (Participants) | 42 | 65 | 0 | 0 | 0 | 0 | 0
  Stage 1 Baseline | 0.080 (0.071) | 0.0755 (0.079) |  |  |  |  |
  Change from Baseline at Week 6: number analyzed (Participants) | 39 | 49 | 0 | 0 | 0 | 0 | 0
  Change from Baseline at Week 6 | -0.021 (0.064) | -0.004 (0.082) |  |  |  |  |
  Stage 2 Baseline: number analyzed (Participants) | 0 | 0 | 17 | 25 | 0 | 0 | 0
  Stage 2 Baseline |  |  | 0.040 (0.049) | 0.071 (0.063) |  |  |
  Change from Baseline at Week 12: number analyzed (Participants) | 0 | 0 | 17 | 25 | 0 | 0 | 0
  Change from Baseline at Week 12 |  |  | 0.000 (0.045) | -0.027 (0.051) |  |  |
Statistical Analysis 1: Comparison: Stage 1: AVP-786 vs Stage 1: Placebo vs Stage 1 Placebo Non-responders; Stage 2: Placebo vs Stage 1 Placebo Non-responders; Stage 2: AVP-786; Test type: Superiority; p = 0.246, ANCOVA; SPCD Weighted OLS z-statistic = -1.159, 95% CI 2-sided [-3.119 to 0.801]

25. Secondary Outcome: Change From Baseline in the EEfRT Score for 50% Probability-Proportion High Effort Opts 1st 50 at Week 6 and Week 12
Description: The EEfRT is a multi-trial computerized test that reliably measures drug effects on the willingness to expend effort in relation to the amount of reward or probability of reward. For each trial, participants are asked to choose between 2 tasks that differ in difficulty level and are associated with varying levels of monetary reward. EEfRT scores are analyzed for 8 variables. Variable 5 is the proportion of hard task choices made for the medium (50%) probability condition during the first 50 trials of the task. Scores range from 0 to 1, with higher scores indicative of greater effort expenditure. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Week 6 (Stage 1); Baseline (Week 6) and Week 12 (Stage 2)
Population: Stage 1 and Stage 2 mITT Populations. Only those participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1: AVP-786 | Stage 1: Placebo | Stage 1 Placebo Non-responders; Stage 2: Placebo | Stage 1 Placebo Non-responders; Stage 2: AVP-786 | Stage 1 Placebo Responders; Stage 2: Placebo | Stage 1 Placebo Responders; Stage 2: AVP-786 | Stage 1 AVP-786; Stage 2: AVP-786
Number analyzed (Participants) | 42 | 65 | 17 | 25 | 0 | 0 | 0
score on a scale
  Stage 1 Baseline: number analyzed (Participants) | 42 | 65 | 0 | 0 | 0 | 0 | 0
  Stage 1 Baseline | 0.088 (0.070) | 0.078 (0.081) |  |  |  |  |
  Change from Baseline at Week 6: number analyzed (Participants) | 39 | 49 | 0 | 0 | 0 | 0 | 0
  Change from Baseline at Week 6 | -0.026 (0.055) | -0.012 (0.102) |  |  |  |  |
  Stage 2 Baseline: number analyzed (Participants) | 0 | 0 | 17 | 25 | 0 | 0 | 0
  Stage 2 Baseline |  |  | 0.060 (0.057) | 0.062 (0.078) |  |  |
  Change from Baseline at Week 12: number analyzed (Participants) | 0 | 0 | 17 | 25 | 0 | 0 | 0
  Change from Baseline at Week 12 |  |  | -0.016 (0.068) | -0.005 (0.083) |  |  |
Statistical Analysis 1: Comparison: Stage 1: AVP-786 vs Stage 1: Placebo vs Stage 1 Placebo Non-responders; Stage 2: Placebo vs Stage 1 Placebo Non-responders; Stage 2: AVP-786; Test type: Superiority; p = 0.818, ANCOVA; SPCD Weighted OLS z-statistic = 0.231, 95% CI 2-sided [-1.729 to 2.191]

26. Secondary Outcome: Change From Baseline in the EEfRT Score for 88% Probability-Proportion High Effort Opts 1st 50 at Week 6 and Week 12
Description: The EEfRT is a multi-trial computerized test that reliably measures drug effects on the willingness to expend effort in relation to the amount of reward or probability of reward. For each trial, participants are asked to choose between 2 tasks that differ in difficulty level and are associated with varying levels of monetary reward. EEfRT scores are analyzed for 8 variables. Variable 6 is the proportion of hard task choices made for the hard (88%) probability condition during the first 50 trials of the task. Scores range from 0 to 1, with higher scores indicative of greater effort expenditure. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Week 6 (Stage 1); Baseline (Week 6) and Week 12 (Stage 2)
Population: Stage 1 and Stage 2 mITT Populations. Only those participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1: AVP-786 | Stage 1: Placebo | Stage 1 Placebo Non-responders; Stage 2: Placebo | Stage 1 Placebo Non-responders; Stage 2: AVP-786 | Stage 1 Placebo Responders; Stage 2: Placebo | Stage 1 Placebo Responders; Stage 2: AVP-786 | Stage 1 AVP-786; Stage 2: AVP-786
Number analyzed (Participants) | 42 | 65 | 17 | 25 | 0 | 0 | 0
score on a scale
  Stage 1 Baseline: number analyzed (Participants) | 42 | 65 | 0 | 0 | 0 | 0 | 0
  Stage 1 Baseline | 0.082 (0.063) | 0.081 (0.086) |  |  |  |  |
  Change from Baseline at Week 6: number analyzed (Participants) | 39 | 49 | 0 | 0 | 0 | 0 | 0
  Change from Baseline at Week 6 | -0.021 (0.072) | -0.006 (0.097) |  |  |  |  |
  Stage 2 Baseline: number analyzed (Participants) | 0 | 0 | 17 | 25 | 0 | 0 | 0
  Stage 2 Baseline |  |  | 0.052 (0.065) | 0.078 (0.074) |  |  |
  Change from Baseline at Week 12: number analyzed (Participants) | 0 | 0 | 17 | 25 | 0 | 0 | 0
  Change from Baseline at Week 12 |  |  | -0.015 (0.047) | -0.015 (0.070) |  |  |
Statistical Analysis 1: Comparison: Stage 1: AVP-786 vs Stage 1: Placebo vs Stage 1 Placebo Non-responders; Stage 2: Placebo vs Stage 1 Placebo Non-responders; Stage 2: AVP-786; Test type: Superiority; p = 0.968, ANCOVA; SPCD Weighted OLS z-statistic = -0.040, 95% CI 2-sided [-2.00 to 1.92]

27. Secondary Outcome: Change From Baseline in the EEfRT Score for All-Proportion High Effort Opts 1st 50 at Week 6 and Week 12
Description: The EEfRT is a multi-trial computerized test that reliably measures drug effects on the willingness to expend effort in relation to the amount of reward or probability of reward. For each trial, participants are asked to choose between 2 tasks that differ in difficulty level and are associated with varying levels of monetary reward. EEfRT scores are analyzed for 8 variables. Variable 7 is the overall proportion of hard task choices made for the first 50 trials of the task. Scores range from 0 to 1, with higher scores indicative of greater effort expenditure. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Week 6 (Stage 1); Baseline (Week 6) and Week 12 (Stage 2)
Population: Stage 1 and Stage 2 mITT Populations. Only those participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1: AVP-786 | Stage 1: Placebo | Stage 1 Placebo Non-responders; Stage 2: Placebo | Stage 1 Placebo Non-responders; Stage 2: AVP-786 | Stage 1 Placebo Responders; Stage 2: Placebo | Stage 1 Placebo Responders; Stage 2: AVP-786 | Stage 1 AVP-786; Stage 2: AVP-786
Number analyzed (Participants) | 42 | 65 | 17 | 25 | 0 | 0 | 0
score on a scale
  Stage 1 Baseline: number analyzed (Participants) | 42 | 65 | 0 | 0 | 0 | 0 | 0
  Stage 1 Baseline | 0.251 (0.185) | 0.234 (0.234) |  |  |  |  |
  Change from Baseline at Week 6: number analyzed (Participants) | 39 | 49 | 0 | 0 | 0 | 0 | 0
  Change from Baseline at Week 6 | -0.068 (0.167) | -0.022 (0.261) |  |  |  |  |
  Stage 2 Baseline: number analyzed (Participants) | 0 | 0 | 17 | 25 | 0 | 0 | 0
  Stage 2 Baseline |  |  | 0.152 (0.161) | 0.210 (0.199) |  |  |
  Change from Baseline at Week 12: number analyzed (Participants) | 0 | 0 | 17 | 25 | 0 | 0 | 0
  Change from Baseline at Week 12 |  |  | -0.032 (0.144) | -0.047 (0.176) |  |  |
Statistical Analysis 1: Comparison: Stage 1: AVP-786 vs Stage 1: Placebo vs Stage 1 Placebo Non-responders; Stage 2: Placebo vs Stage 1 Placebo Non-responders; Stage 2: AVP-786; Test type: Superiority; p = 0.760, ANCOVA; SPCD Weighted OLS z-statistic = -0.306, 95% CI 2-sided [-2.266 to 1.654]

28. Secondary Outcome: Change From Baseline in the EEfRT Score for Difference - Proportion High Effort Opts 1st 50 at Week 6 and Week 12
Description: The EEfRT is a multi-trial computerized test that reliably measures drug effects on the willingness to expend effort in relation to the amount of reward or probability of reward. For each trial, participants are asked to choose between 2 tasks that differ in difficulty level and are associated with varying levels of monetary reward. EEfRT scores are analyzed for 8 variables. Variable 8 is the difference between the proportion of hard task choices made for the high probability condition during the first 50 trials of the task. Scores range from -1 to 1, with higher scores indicative of greater sensitivity to probability information. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Week 6 (Stage 1); Baseline (Week 6) and Week 12 (Stage 2)
Population: Stage 1 and Stage 2 mITT Populations. Only those participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1: AVP-786 | Stage 1: Placebo | Stage 1 Placebo Non-responders; Stage 2: Placebo | Stage 1 Placebo Non-responders; Stage 2: AVP-786 | Stage 1 Placebo Responders; Stage 2: Placebo | Stage 1 Placebo Responders; Stage 2: AVP-786 | Stage 1 AVP-786; Stage 2: AVP-786
Number analyzed (Participants) | 42 | 65 | 17 | 25 | 0 | 0 | 0
score on a scale
  Stage 1 Baseline: number analyzed (Participants) | 42 | 65 | 0 | 0 | 0 | 0 | 0
  Stage 1 Baseline | 0.002 (0.041) | 0.006 (0.037) |  |  |  |  |
  Change from Baseline at Week 6: number analyzed (Participants) | 39 | 49 | 0 | 0 | 0 | 0 | 0
  Change from Baseline at Week 6 | -0.001 (0.054) | -0.002 (0.050) |  |  |  |  |
  Stage 2 Baseline: number analyzed (Participants) | 0 | 0 | 17 | 25 | 0 | 0 | 0
  Stage 2 Baseline |  |  | 0.012 (0.032) | 0.006 (0.034) |  |  |
  Change from Baseline at Week 12: number analyzed (Participants) | 0 | 0 | 17 | 25 | 0 | 0 | 0
  Change from Baseline at Week 12 |  |  | -0.015 (0.037) | 0.012 (0.039) |  |  |
Statistical Analysis 1: Comparison: Stage 1: AVP-786 vs Stage 1: Placebo vs Stage 1 Placebo Non-responders; Stage 2: Placebo vs Stage 1 Placebo Non-responders; Stage 2: AVP-786; Test type: Superiority; p = 0.214, ANCOVA; SPCD Weighted OLS z-statistic = 1.243, 95% CI 2-sided [-0.717 to 3.203]

29. Secondary Outcome: Number of Participants With a Reduction of 20% or Greater in the PANSS Total Score at Week 6 and Week 12
Description: Treatment effect was evaluated by analyzing the proportion of participants with a 20% reduction from Baseline in the PANSS total score with SPCD analysis.
Time Frame: Baseline and Week 6 (Stage 1); Baseline (Week 6) and Week 12 (Stage 2)
Population: Stage 1 and Stage 2 mITT Populations
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1: AVP-786 | Stage 1: Placebo | Stage 1 Placebo Non-responders; Stage 2: Placebo | Stage 1 Placebo Non-responders; Stage 2: AVP-786 | Stage 1 Placebo Responders; Stage 2: Placebo | Stage 1 Placebo Responders; Stage 2: AVP-786 | Stage 1 AVP-786; Stage 2: AVP-786
Number analyzed (Participants) | 47 | 80 | 30 | 33 | 0 | 0 | 0
Participants
  Week 6; Response = Yes: number analyzed (Participants) | 47 | 80 | 0 | 0 | 0 | 0 | 0
  Week 6; Response = Yes | 5 | 3 |  |  |  |  |
  Week 6; Response = No: number analyzed (Participants) | 47 | 80 | 0 | 0 | 0 | 0 | 0
  Week 6; Response = No | 42 | 77 |  |  |  |  |
  Week 12; Response = Yes: number analyzed (Participants) | 0 | 0 | 30 | 33 | 0 | 0 | 0
  Week 12; Response = Yes |  |  | 1 | 3 |  |  |
  Week 12; Response = No: number analyzed (Participants) | 0 | 0 | 30 | 33 | 0 | 0 | 0
  Week 12; Response = No |  |  | 29 | 30 |  |  |
Statistical Analysis 1: Comparison: Stage 1: AVP-786 vs Stage 1: Placebo vs Stage 1 Placebo Non-responders; Stage 2: Placebo vs Stage 1 Placebo Non-responders; Stage 2: AVP-786; Test type: Superiority; p = 0.071, SPCD 1 degree of freedom score test

30. Secondary Outcome: Change From Baseline in the 4-Item NSA (NSA-4) Total Score at Week 6 and Week 12
Description: The NSA-4 is comprised of the 4 NSA-16 items as follows: 1) restricted speech quantity, 2) emotion: reduced range, 3) reduced social drive, and 4) reduced interests, as well as an overall global rating of negative symptoms. The NSA-16 is a measure of the presence, severity, and range of negative symptoms associated with schizophrenia. It has a high interrater and test-retest reliability across languages and cultures. The possible NSA-4 total score ranges from 4 to 24, with higher scores indicating greater clinical severity of symptoms. Change was Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Week 6 (Stage 1); Baseline (Week 6) and Week 12 (Stage 2)
Population: Stage 1 and Stage 2 mITT Populations. Only those participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1: AVP-786 | Stage 1: Placebo | Stage 1 Placebo Non-responders; Stage 2: Placebo | Stage 1 Placebo Non-responders; Stage 2: AVP-786 | Stage 1 Placebo Responders; Stage 2: Placebo | Stage 1 Placebo Responders; Stage 2: AVP-786 | Stage 1 AVP-786; Stage 2: AVP-786
Number analyzed (Participants) | 47 | 80 | 30 | 33 | 0 | 0 | 0
score on a scale
  Stage 1 Baseline: number analyzed (Participants) | 47 | 80 | 0 | 0 | 0 | 0 | 0
  Stage 1 Baseline | 17.4 (2.44) | 17.3 (2.36) |  |  |  |  |
  Change from Baseline at Week 6: number analyzed (Participants) | 47 | 70 | 0 | 0 | 0 | 0 | 0
  Change from Baseline at Week 6 | -1.0 (2.10) | -1.0 (1.92) |  |  |  |  |
  Stage 2 Baseline: number analyzed (Participants) | 0 | 0 | 30 | 33 | 0 | 0 | 0
  Stage 2 Baseline |  |  | 16.5 (2.64) | 16.4 (2.84) |  |  |
  Change from Baseline at Week 12: number analyzed (Participants) | 0 | 0 | 29 | 32 | 0 | 0 | 0
  Change from Baseline at Week 12 |  |  | -0.5 (2.01) | -0.5 (1.93) |  |  |
Statistical Analysis 1: Comparison: Stage 1: AVP-786 vs Stage 1: Placebo vs Stage 1 Placebo Non-responders; Stage 2: Placebo vs Stage 1 Placebo Non-responders; Stage 2: AVP-786; Treatment differences in each stage were estimated by the MMRM; Test type: Superiority; p = -0.06, Mixed Models Analysis; SPCD Weighted OLS z-statistic = 0.951, 95% CI 2-sided [-1.009 to 2.911]

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) were collected for approximately 90 days.
Description: Treatment-emergent adverse events (TEAEs) are reported and defined as any AE that first occurred, or worsened, after the first dose of study medication and within 30 days after the permanent discontinuation of study medication (first dose on or before AE start date which was on or before the date of last dose +30 days). All serious adverse events are reported.
Groups:
- All Placebo: Participants who received placebo in Stage 1 or Stage 2.
- All AVP-786: Participants who received AVP-786 in Stage 1 or Stage 2 (up to a target dose of AVP-786-34/4.9 milligrams twice a day [d6-DM 34 mg/Q 4.9 mg BID]).
Arm/Group | All Placebo | All AVP-786
All-Cause Mortality (participants affected / at risk) | 0/96 | 0/88
Serious Adverse Events (participants affected / at risk) | 2/96 | 0/88
Other Adverse Events (participants affected / at risk) | 39/96 | 30/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Placebo (N=96) | All AVP-786 (N=88)
Urinary tract infection (Infections and infestations) | 1 | 0
Schizophrenia (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Placebo (N=96) | All AVP-786 (N=88)
Dry mouth (Gastrointestinal disorders) | 1 | 4
Diarrhoea (Gastrointestinal disorders) | 3 | 2
Glossitis (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Dental discomfort (Gastrointestinal disorders) | 1 | 0
Dizziness (Nervous system disorders) | 3 | 3
Headache (Nervous system disorders) | 5 | 2
Paraesthesia (Nervous system disorders) | 1 | 1
Somnolence (Nervous system disorders) | 3 | 1
Dysgeusia (Nervous system disorders) | 1 | 0
Dyskinesia (Nervous system disorders) | 1 | 0
Sedation (Nervous system disorders) | 2 | 0
Syncope (Nervous system disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 4 | 3
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Groin infection (Infections and infestations) | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 1 | 1
Bacterial vaginosis (Infections and infestations) | 0 | 1
Otitis externa (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Conjunctivitis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 2
Blood prolactin increased (Investigations) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Paranoia (Psychiatric disorders) | 1 | 0
Schizophrenia (Psychiatric disorders) | 1 | 0
Vision blurred (Eye disorders) | 0 | 2
Eye pain (Eye disorders) | 1 | 0
Glycosuria (Renal and urinary disorders) | 0 | 1
Urine abnormality (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Scratch (Injury, poisoning and procedural complications) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Fatigue (General disorders) | 2 | 1
Pyrexia (General disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-08-15): https://cdn.clinicaltrials.gov/large-docs/70/NCT02477670/SAP_000.pdf
  • Study Protocol (2016-01-25): https://cdn.clinicaltrials.gov/large-docs/70/NCT02477670/Prot_001.pdf